CLINICAL TRIAL: NCT05742048
Title: Diagnostic Performance of Ultrasound for Primary Survey of Traumatic Long Bone Fractures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelbaky Abdelrahman, Clinical Professor, Assiut University
Other Study IDs: Long bone sonography
Record Dates: First submitted 2023-01-30; First posted 2023-02-23 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-01

CONDITIONS: Trauma
Keywords: Long bone fractures; Bone sonography; Ultrasound Bone scan
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- traumatic patient suspect to have long bone fracture between 18 - 65 years old
  Interventions: Diagnostic Test: traumatic patient suspect to have long bone fracture between 18 - 65 years old

INTERVENTIONS:
Diagnostic Test: traumatic patient suspect to have long bone fracture between 18 - 65 years old — Number of patients diagnosed to have a long bone fracture by using ultrasound. Number of patients diagnosed to have a long bone fracture by using x-ray . Comparison between Ultrasound bone scan result and X-ray imaging accuracy and sensitivity.

SUMMARY:
Long bone fractures are among the most traumatic patients seen in emergency departments. Using ultrasound to diagnose long bone fractures can reduce the risk of complications occurring During the primary and secondary survey.

The diagnosis of long bone fractures is traditionally accomplished through plain radiographs taken at perpendicular angles to each other.

Because of the resources required for radiographic capability, X-ray can be inaccessible in rural or remote areas, or in hospital during break time, In settings where a radiography technologist is not present on-site or in patient have conditions do for him limitations movement Using ultrasound machines to do patient examination can be performed earlier of assessment, and at the bedside, reducing diagnostic delays and time to initiation of management. Additional Advantages of Ultrasound include its simplicity, portability, repeatability, and its lack of ionizing radiation. Using ultrasound technology don't need equipment for lead protectors on health care providers, as well as the harmful effects to patients of ionizing radiation and safe to use with pregnant patients in the first and second trimester.

However, this technique can be impractical because the training necessary for the use of this technology Diagnosis of long bone fractures in primary assessment can decrease risk of complications such as shock, bleeding, swelling, embolism compartment syndrome, vascular or neurological damage and patient's transposition related change shape and type of a fracture. that complications can lead to life-threatening conditions up to death specifically in geriatric and paediatric Patients

DETAILED DESCRIPTION:
Primary assessment for traumatic patient included:

A- Airway with cervical spine precautions /or protection: This assessment is of the patency of the patient's airway.

B- Breathing and Ventilation: This assessment is performed first by inspection. C- circulation with hemorrhage control: Adequate circulation is required for oxygenation to the brain and other vital organs. Blood loss is the most common cause of shock in trauma patients.

D- Disability (assessing neurological status): A rapid assessment of the patient's neurologic status is necessary on arrival in the emergency department.

E- Exposure and Environmental Control: The patient should be completely undressed and exposed to ensure no injuries are missed.

Adjuncts to the Primary Survey:After the ABCDEs of the primary survey, several adjuncts assist in the evaluation of other life-threatening processes:

ECG Urinary Catheters Gastric catheters FAST Examination:"Focused Assessment with Sonography in Trauma"

Long bone ultrasound scan:

To exclude risk of harm from long bone fractures, do Examination of the upper and lower extremities to verify direct hit or fall within have evidence of pain, tenderness, redness, swelling or any sign of trauma on the patient's extremities? After identifying the suspected suffering places, The ultrasound probe placed the lateral surface of the bone transversely and longitudinally, and the cortex section is examined.

First, the probe placement transversely onto the surface of the bone to examine the presence of skip.

Longitudinal and transverse scans should be coupled in each patient to confirm the focal interruption of the hyperechoic cortical bone. The longitudinal scan allows a panoramic view of the cortical irregularity while the transverse scan often guarantees a better visualization of the shift/rotation of the pathological bony fragment Bone fractures can be visualized as a cortical contour interruption, imaging also allows the identification of surrounding hematoma and the evaluation of bone callus during its different phases In the next step (secondary survey), standard bone radiography x-ray will be performed, anteroposterior and lateral to compare between the results.

After bone sonography scan in patients suspected to have upper and lower limb trauma, The Ultrasound probe will be placed over the area of maximum pain to find any abnormality suspected in soft tissue, vascular supplies, muscle and tendon health.

2.4.5 -Research outcome measures:

a. Primary (main): Number of patients diagnosed to have a long bone fracture by using ultrasound. Number of patients diagnosed to have a long bone fracture by using x-ray . Comparison between Ultrasound bone scan result and X-ray imaging accuracy and sensitivity.

Secondary (subsidiary):

The skin, soft tissue, and most parts of the musculoskeletal system are relatively the superficial anatomical structures it's ideal targets for ultrasound examination, Such as soft tissue abnormalities, vascularity and muscle state in traumatic patients. Distinguishing flexibility positioning of the part without making the patient too uncomfortable adds to the list advantages of this modality.

ELIGIBILITY:
Inclusion Criteria:

* traumatic patient suspect to have long bone fracture between 18 - 65 years old

Exclusion Criteria:

* Patient refused to participate in the research.
* Previously diagnosed patient with long bone fractures.
* Critically injured patients
* Obese patient (BMI) > 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic patient between 18 - 60 years old suspect to have long bone fracture with in the first 24 hours from trauma
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between Ultrasound bone scan result and X-ray imaging accuracy and sensitivity. | through study completion, an average of 1 year
  measure of sensitivity, specificity, positive and negative predictive values and accuracy of ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] O'Brien AJ, Moussa MA. Using ultrasound to diagnose long bone fractures. JAAPA. 2020 Feb;33(2):33-37. doi: 10.1097/01.JAA.0000651736.02537.ef. PMID 31990832
- [Result] Nicholson JA, Makaram N, Simpson A, Keating JF. Fracture nonunion in long bones: A literature review of risk factors and surgical management. Injury. 2021 Jun;52 Suppl 2:S3-S11. doi: 10.1016/j.injury.2020.11.029. Epub 2020 Nov 11. PMID 33221036
- [Result] Chartier LB, Bosco L, Lapointe-Shaw L, Chenkin J. Use of point-of-care ultrasound in long bone fractures: a systematic review and meta-analysis. CJEM. 2017 Mar;19(2):131-142. doi: 10.1017/cem.2016.397. Epub 2016 Dec 5. PMID 27916021
- [Result] Gharahbaghian L, Anderson KL, Lobo V, Huang RW, Poffenberger CM, Nguyen PD. Point-of-Care Ultrasound in Austere Environments: A Complete Review of Its Utilization, Pitfalls, and Technique for Common Applications in Austere Settings. Emerg Med Clin North Am. 2017 May;35(2):409-441. doi: 10.1016/j.emc.2016.12.007. PMID 28411935
- See also: Use of point-of-care ultrasound in long bone fractures: a systematic review and meta-analysis Lucas B Chartier et al. CJEM. 2017 Mar. — https://pubmed.ncbi.nlm.nih.gov/27916021/
- See also: Mitchell C. World Radiography Day: two-thirds of the world's population has no access to diagnostic imaging, — http://www.paho.org/hq/index.php?option=com_content&view=